CLINICAL TRIAL: NCT01079390
Title: An Acupuncture fMRI Study on Chronic Pain: Response Reliability and Dose Effect
Brief Title: An Acupuncture Functional Magnetic Resonance Imaging (fMRI) Study on Chronic Pain: Response Reliability and Dose Effect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jian Kong, Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2009-P-000904; 1R21AT004497-01A2 (NIH)
Record Dates: First submitted 2010-03-01; First posted 2010-03-03 (Estimated); Results first posted 2017-08-10 (Actual); Last update posted 2017-08-10 (Actual); Status verified 2017-02

CONDITIONS: Osteoarthritis, Knee
Keywords: acupuncture; osteoarthritis; fMRI
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High dose acupuncture (Experimental): six needle applied during acupuncture
  Interventions: Device: acupuncture
- Low dose acupuncture (Experimental): two needles will be applied.
  Interventions: Device: acupuncture
- placebo acupuncture (Placebo Comparator): sham acupuncture treatment will be applied
  Interventions: Device: acupuncture

INTERVENTIONS:
Device: acupuncture — patient will receive high dose, low dose or sham acupuncture treatment.

SUMMARY:
In this proposal, we plan to dynamically investigate brain response to verum acupuncture (of two different "doses") and placebo acupuncture, using a paradigm that approximates clinical acupuncture practice across multiple treatment sessions in knee osteoarthritis (OA) patients. This proposal aims to: 1) characterize session-to-session brain responses to verum / sham acupuncture treatment (reliability of response) for OA patients, and 2) investigate how different "doses" of acupuncture influence brain response and acupuncture efficacy (impact of dose). The findings of this project will deepen our biological understanding on why and how acupuncture can treat chronic pain and what happens in the brain during the multiple-session acupuncture treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers 40-70 years of age.
2. Meet the Classification Criteria of the American College of Rheumatology for osteoarthritis of the left / right knee for at least the past 3 months, as determined by the referring physician.
3. Radiographic evidence of Grade 2 or 3 knee OA using the Kellgren-Lawrence Scale [78, 85-87].
4. Patients must have moderate or greater clinically significant pain on most days during the past month (more than 15 days out of 30, of average daily pain of >3/10) in the left or right knee.
5. At least a 10th grade English-reading level; English can be a second language provided that the patients feel they understand all the questions used in the assessment measures.

Exclusion Criteria:

1. Any interventional procedure for knee pain, including corticosteroid injections (within 6 months, [88]) to the knee.
2. Prior acupuncture treatment for any condition. Because we are using a placebo needle as a control, acupuncture-naive patients are necessary to maximize the benefits of blinding and to control expectancy.
3. The intent to undergo surgery during the time of involvement in the study.
4. Presence of any illness or medication use that is judged to interfere with the trial. For example: skin irritations around the knee such as psoriasis; bleeding disorders or anticoagulant use that would be contraindications for acupuncture; opioids or benzodiazepines, which may alter pain sensitivity and BOLD response.
5. Knee pain due to other causes, such as inflammation or malignancy, other pain disorders that may refer pain to the leg, OA of ipsilateral hip, diagnosis of RA.
6. Non-ambulatory status.
7. History of cardiac, respiratory, or nervous system disease that, in the investigator's judgment, precludes participation in the study because of a heightened potential for adverse outcome. For example: asthma or claustrophobia.
8. Presence of any contraindications to fMRI scanning. For example: cardiac pacemaker, metal implants, fear of closed spaces, pregnancy.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-01; Primary Completion 2013-01 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jian Kong, Principal Investigator — Massachusetts General Hosptial
Locations (1):
- Massachusetts General Hosptial, Charlestown, Massachusetts, United States

REFERENCES:
- [Derived] Chen X, Spaeth RB, Freeman SG, Scarborough DM, Hashmi JA, Wey HY, Egorova N, Vangel M, Mao J, Wasan AD, Edwards RR, Gollub RL, Kong J. The modulation effect of longitudinal acupuncture on resting state functional connectivity in knee osteoarthritis patients. Mol Pain. 2015 Oct 29;11:67. doi: 10.1186/s12990-015-0071-9. PMID 26511911
- [Derived] Chen X, Spaeth RB, Retzepi K, Ott D, Kong J. Acupuncture modulates cortical thickness and functional connectivity in knee osteoarthritis patients. Sci Rep. 2014 Sep 26;4:6482. doi: 10.1038/srep06482. PMID 25258037

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty-four acupuncture naïve patients aged 43-70 with a diagnosis of chronic osteoarthritis in the right and/or left knee participated in the study. 30 (13 females) completed all study procedures. Fourteen subjects did not complete the study. All subjects were recruited form the Boston area over the course of the past 3 years.
Pre-assignment Details: Fourteen subjects did not complete the study due to problems with scheduling (6), ineligibility at screening (3), disinterest (2), claustrophobia (1), or inability to adhere to study requirements in scanner (2). Of the 14 subjects who dropped, four dropped out after randomization.
Groups:
- High Dose Acupuncture: six needle applied during acupuncture
  acupuncture : patient will receive high dose, low dose or sham acupuncture treatment.
- Low Dose Acupuncture: two needles will be applied.
  acupuncture : patient will receive high dose, low dose or sham acupuncture treatment.
- Placebo Acupuncture: sham acupuncture treatment will be applied
  acupuncture : patient will receive high dose, low dose or sham acupuncture treatment.
Period: Overall Study
Arm/Group | High Dose Acupuncture | Low Dose Acupuncture | Placebo Acupuncture
Started | 15 | 15 | 14
Completed | 10 | 10 | 10
Not Completed | 5 | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose Acupuncture | Low Dose Acupuncture | Placebo Acupuncture | Total
Number analyzed (Participants) | 15 | 15 | 14 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 14 | 44
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (9) | 58 (8) | 54 (7) | 58 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 4 | 17
  Male | 10 | 7 | 10 | 27
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 14 | 44

OUTCOME MEASURES:

1. Primary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS Pain Rating) at 5-7 Weeks Post-Treatment
Description: The Knee injury and Osteoarthritis Outcome Score (KOOS) was used to measure clinical outcomes. KOOS is measured on a scale from 0-4 with 0 being no pain and 4 being extreme pain (the worst). The KOOS is comprised of 5 subscales, each of which produces an outcome score. These subscales include pain, other symptoms, function in daily living (ADL), function in sport and recreation, and knee-related quality of life (QOL). Based on previous studies, subscale scores of the KOOS related to pain, function in daily living, and function in sport and recreation were selected as the primary outcome of the present study. For each subscale, a normalized score was calculated, where 0 indicated the most extreme symptoms/pain and 100 indicated no symptoms/pain.
Time Frame: One post-treatment measurement 5-7 weeks after baseline
Measure: Mean (Standard Deviation); unit: units on KOOS scale
Arm/Group | High Dose Acupuncture | Low Dose Acupuncture | Placebo Acupuncture
Number analyzed (Participants) | 10 | 10 | 10
units on KOOS scale | 59 (13) | 53 (9) | 56 (19)

2. Primary Outcome: Cortical Thickness Changes at 5-7 Weeks Post-Treatment
Description: All eligible patients were scanned using fMRI while receiving treatment during acupuncture sessions 1, 3, and 6. Structural MRI data were only compared between Session 1 (pre-treatment) and Session 6 (post-treatment). The structural data was analyzed using FreeSurfer software.
Time Frame: 2 days; one at baseline and another post-treatment measurement taken 5-7 weeks after baseline
Population: We combined low and high dose acupuncture into one group because we found there were not clinical differences between the two group.
Measure: Mean (Standard Deviation); unit: millimeters
Groups:
- Acupuncture: six needle applied during acupuncture
  acupuncture : patient will receive high or low dose.
- Placebo Acupuncture: sham acupuncture treatment will be applied
  acupuncture : patient will receive sham acupuncture treatment.
Arm/Group | Acupuncture | Placebo Acupuncture
Number analyzed (Participants) | 20 | 10
millimeters | 2.9 (0.15) | 3.13 (0.28)

ADVERSE EVENTS:
Arm/Group | High Dose Acupuncture | Low Dose Acupuncture | Placebo Acupuncture
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/14

LIMITATIONS AND CAVEATS:
Limitations of the study are the small sample size as well as the effects of factors such as age, gender, and chronic duration of pain.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No